CLINICAL TRIAL: NCT05932589
Title: Characterization of Translatable Neurophysiological Biomarkers to Enhance Therapeutic Development in Rett Syndrome
Brief Title: Neurophysiologic Biomarkers in Rett Syndrome
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 22-020633; 1R61NS130216-01 (NIH)
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Rett Syndrome; RTT; Rett Syndrome, Atypical
Keywords: Biomarker; EEG; Evoked Potentials; MECP2
MeSH Terms: conditions — Rett Syndrome; Rett Syndrome, Atypical | interventions — Evoked Potentials, Visual; asparaginylendopeptidase

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RTT Females: Females with Rett Syndrome
  Interventions: Other: EEG and Auditory and Visual Evoked Potentials (AEP and VEP); Other: Clinical assessment
- Controls: Females with typical development
  Interventions: Other: EEG and Auditory and Visual Evoked Potentials (AEP and VEP)

INTERVENTIONS:
Other: EEG and Auditory and Visual Evoked Potentials (AEP and VEP) — Through up to eight standardized sessions, participants will undergo AEP and VEP, as well as resting state EEG.
Other: Clinical assessment — Established clinical measures for RTT will be collected for RTT participants
  Groups: RTT Females

SUMMARY:
The goal of this observational study is to identify candidate biomarkers in individuals with Rett Syndrome (RTT). The main questions it aims to answer are:

* Do these biomarkers change during clinical changes in individuals with RTT?
* Are biomarkers stable over time in clinically stable individuals?
* Do these biomarkers correlate with severity of RTT?

Participants will be asked to undergo an electroencephalogram (EEG) with measurements of Evoked Potentials (EP) to measure electrical activity in the brain.

Researchers will compare findings in individuals with RTT to those in typically developing individuals to see if there are differences between the two groups.

DETAILED DESCRIPTION:
The main goal of the project is to identify potential biomarkers that can become measures for intervention and other translational studies and, at the same time, provide insight into abnormal synaptic activity and pathogenesis of RTT. Therefore, the proposed assessments will be performed with females with RTT and age matched typically developing females. These electrophysiological assessments will be compared to established clinical outcome measures from previous work in the NIH funded Rett and Rett related disorders natural history study. The neurophysiological parameters for RTT will be correlated with each other and also to disease staging, overall clinical severity scores and through exploratory analyses with specific clinical features. The investigators will also be testing procedures to perform the recordings, electrode types and placement, and ways to reduce movement and artifact within the data to establish best practices.

ELIGIBILITY:
Inclusion Criteria:

1. Rett Group: Females ages 3-18 (inclusive) with a clinical diagnosis of RTT with a likely pathogenic or known pathogenic variant in MECP2.
2. Likely Rett Group: Females from 1 year to < 5 years of age with MECP2 variant if regression has not yet occurred or child is within 6 months of last skill loss.
3. Typically developing (TD) Group: Females age matched to RTT population (1-18) with no developmental or cognitive concerns as assessed using the Child/Adult Behavioral Checklist, Survey of Well-Being of Young Children (<5yo), or the Wide Range Achievement Test-4 (>5 yo).

Exclusion Criteria:

Rett and Likely Rett Groups:

1. Presence of a duplication in MECP2 or any other identified pathogenic mutation in another gene.
2. Active medical conditions not typically found in RTT.

Typically Developing Group:

1. Score below norms on the performance tests
2. Have a known neurological disorder (excluding migraine)
3. Being on neuroactive medications.

Ages: 1 Year to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Enrolled participants with Rett syndrome will include individuals receiving clinical care through the Rett Syndrome clinics at participating sites. Typically developing individuals will be recruited using study recruitment centers or family members of Rett participants at each site. Each of the sites are International Rett Syndrome Foundation Centers of Excellence (Rettsyndrome.org).
Sampling Method: Non-Probability Sample
Enrollment: 202 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Auditory Evoked Potential (AEP) latency (ms) | 5 years
  Calculated N1, P1 latencies in Cz and other electrodes [posterior temporal region (T5/P3/T3) electrodes], will be used for analysis.
Auditory Evoked Potential (AEP) amplitude | 5 years
  Amplitude of P1, P2 and N1 peaks (uV)
Visual Evoked Potential (VEP) latencies (ms) | 5 years
  The latencies of the N1, P1, and N2 components will be identified primarily at occipital electrodes with Oz will be the primary electrode of analysis. N1-P1 time will be analyzed.
Visual Evoked Potential (VEP) amplitude | 5 years
  N1-P1 amplitude at Oz and other occipital electrodes will be calculated.
EEG Analysis | 5 years
  EEG Root mean square (RMS) amplitude, Amplitude variability, 1/f constant, power bands in typical bands (Delta, theta, alpha, Beta, gamma) and ratios will be calculated.

SECONDARY OUTCOMES:
AEP spectral analysis, dipole determination and spatial distribution | 5 years
  spectral analysis of the individual waveforms, dipole determination of N1 and P1 peaks and spatial distribution of peak values.
VEP spectral analysis, dipole determination and spatial distribution | 5 years
  spectral analysis of the individual waveforms, dipole determination of N1 and P1 peaks and spatial distribution of peak values.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Marsh, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia; Jeffrey Neul, MD, PhD, Principal Investigator — Vanderbilt University Medical Cener
Locations (6):
- United States (6):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Boston Children's Hospital, Brookline, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The investigators intend to submit deidentified patient data into the National Database for Autism Research (NDAR) and database of Genotypes and Phenotypes (dbGaP). Study protocols and data analysis methods will be shared through future publications.
Time Frame: Available data from this observational study will be released to the repository and will become available to the scientific community one year after publication of planned analyses, or after a period of 5 years from the date when the data were collected, whichever comes first.
Access Criteria: National Institute of Mental Health (NIMH) Data Archive (NDA) policy will govern access criteria.

REFERENCES:
- [Background] Saby JN, Peters SU, Roberts TPL, Nelson CA, Marsh ED. Evoked Potentials and EEG Analysis in Rett Syndrome and Related Developmental Encephalopathies: Towards a Biomarker for Translational Research. Front Integr Neurosci. 2020 May 28;14:30. doi: 10.3389/fnint.2020.00030. eCollection 2020. PMID 32547374
- [Background] Saby JN, Benke TA, Peters SU, Standridge SM, Matsuzaki J, Cutri-French C, Swanson LC, Lieberman DN, Key AP, Percy AK, Neul JL, Nelson CA, Roberts TPL, Marsh ED. Multisite Study of Evoked Potentials in Rett Syndrome. Ann Neurol. 2021 Apr;89(4):790-802. doi: 10.1002/ana.26029. Epub 2021 Feb 4. PMID 33480039
- [Background] LeBlanc JJ, DeGregorio G, Centofante E, Vogel-Farley VK, Barnes K, Kaufmann WE, Fagiolini M, Nelson CA. Visual evoked potentials detect cortical processing deficits in Rett syndrome. Ann Neurol. 2015 Nov;78(5):775-86. doi: 10.1002/ana.24513. Epub 2015 Sep 18. PMID 26332183